CLINICAL TRIAL: NCT07188610
Title: PA3-17 Injection for the Treatment of Subjects With Relapsed/Refractory T-Lymphoblastic Leukemia/Lymphoma: A Single-Arm, Open-Label Phase II Clinical Trial
Brief Title: PA3-17 Injection in Adult Patients With CD7-positive Relapsed/Refractory T-lymphoblastic Leukemia/Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-002
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: CD7-positive Relapsed/Refractory T Lymphoblastic Leukemia/Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T cell injection targeting CD7 chimeric antigen receptor (Experimental)
  Interventions: Biological: T cell injection targeting CD7 chimeric antigen receptor

INTERVENTIONS:
Biological: T cell injection targeting CD7 chimeric antigen receptor — After signing the informed consent form, eligible subjects will undergo a single nucleated cell collection for the preparation of CAR-T cells, followed by lymphodepletion pretreatment and a single infusion of PA3-17 injection.

SUMMARY:
**Translation:**

This clinical trial is designed as a single-arm, open-label, multicenter study. After signing the informed consent form, eligible subjects will undergo a single nucleated cell collection for the preparation of CAR-T cells. Following lymphodepletion pretreatment, a single infusion of PA3-17 injection will be administered. Blood samples will be collected from the subjects before and after the infusion for pharmacokinetic, pharmacodynamic, immunogenicity, and safety evaluations. In addition to the baseline period, the treatment phase will involve efficacy assessments at 4 weeks, 2 months, 3 months, and every 3 months thereafter, up to 24 months post-cell infusion. Tumor assessments will continue until disease progression (PD), initiation of new antitumor treatment, death, unacceptable toxicity, investigator decision, or subject's voluntary withdrawal, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Gender: ≥18 years old (inclusive), regardless of gender.
2. Survival Expectancy: ≥3 months.
3. Performance Status: ECOG score 0-1.
4. Diagnosis: Confirmed acute T-cell lymphoblastic leukemia/lymphoma (T-ALL/LBL) according to the WHO fifth edition of the "Classification of Hematopoietic and Lymphoid Tumors," including early T-cell precursor (ETP).
5. Recurrent or Refractory Disease: Subjects with recurrent/refractory T-ALL/LBL (including ETP-ALL/LBL).
6. Screening: Abnormal cells CD7 expression positive.
7. Lesion Assessment: If the subject has only extramedullary lesions, they must have evaluable lesions.
8. Meet the requirements of liver, kidney, heart, and lung functions.
9. No Severe Mental Disorders.
10. Informed Consent: Ability to understand the trial and signed informed consent form.

Exclusion Criteria:

1. Known to have active or uncontrolled autoimmune diseases;
2. Presence of GvHD;
3. History of malignant tumors other than T-ALL/LBL within the past 5 years, except for adequately treated cervical intraepithelial neoplasia, basal cell or squamous cell skin cancer, locally treated prostate cancer, and ductal carcinoma in situ of the breast after radical surgery;
4. Positive test results for hepatitis B, hepatitis C, syphilis, etc.;
5. Severe heart disease;
6. Unstable systemic diseases as judged by the investigator;
7. Presence of active infection or uncontrollable infection requiring systemic treatment;
8. Pregnant or breastfeeding women, and female subjects planning to conceive within 2 years after cell infusion, or male subjects whose partners plan to conceive within 2 years after cell infusion;
9. Subjects who have received CAR-T therapy or other gene-modified cell therapy before screening;
10. Participation in other clinical studies within 1 month before screening (end date of the last application of unapproved innovative drugs);
11. Evidence of central nervous system involvement at the time of subject screening;
12. Situations judged by the investigator as not suitable for cell preparation;
13. Other circumstances deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy | Three months
  Three-month Objective Response Rate (ORR): Proportion of Composite Complete Response Rate (CRc: CR, CRh, CRi, MLFS) and PR

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, Guangdong
  - The First Hospital of Harbin, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Tongji Hospital, Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University (WCHSU), Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No